CLINICAL TRIAL: NCT00645463
Title: A Phase 1, Randomized, Fixed Sequence Study To Evaluate The Effect Of Multiple Dose Administration Of Modified Release Diltiazem On The Multiple Dose Pharmacokinetics Of CP-945,598 In Healthy Overweight And Obese Subjects
Brief Title: Effect of Diltiazem Administration on CP-945,598 Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A5351043
Record Dates: First submitted 2008-03-21; First posted 2008-03-27 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2008-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: CP-945,598
- Group B (Experimental)
  Interventions: Drug: CP-945,598

INTERVENTIONS:
Drug: CP-945,598 — 20 mg CP-945,598 + 240 mg MR Diltiazem
  Arms: Group A
Drug: CP-945,598 — 20 mg CP-945,598 alone
  Arms: Group B

SUMMARY:
A recently completed clinical drug interaction study of CP-945,598 with ketoconazole, a potent CYP3A inhibitor, showed that coadministration of CP-945,598 with ketoconazole results in an approximately 5-fold increase in CP-945,598 total exposure (AUC) and 4-fold increase in Cmax. Therefore, the sensitivity of CP-945,598 pharmacokinetics (PK) to less potent CYP3A inhibitors needs to be characterized to support labeling and registration.

Diltiazem is a known substrate and moderate mechanism-based inhibitor of the CYP3A enzyme system and was chosen as the moderate CYP3A inhibitor for this study as it is a clinically relevant medication likely to be prescribed concomitantly with CP-945,598 given the increased risk of hypertension and cardiovascular disease in the obese patient population.

ELIGIBILITY:
Inclusion Criteria:

* No clinically relevant abnormalities based upon medical history, physical exam, 12-lead ECG, and clinical lab tests
* Body Mass Index (BMI) ~ 27-40 kg/m2, inclusive
* Personally signed inform consent document

Exclusion Criteria:

* Evidence or history of significant acute or chronic disease
* Pregnant or nursing females
* Screening PR interval > 220 msec
* Sitting blood pressure <= 90 mmHg systolic or <= 60 mmHg diastolic

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2007-03; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of CP-945,598 and its metabolite, CE-156,706, (AUCtau, Cmax and Tmax) | Days 7 and 28
Safety endpoints including adverse event monitoring, physical examinations, vital signs, ECGs, and clinical laboratory tests. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Ann Arbor, Michigan, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5351043&StudyName=Effect%20of%20Diltiazem%20Administration%20on%20CP-945%2C598%20Pharmacokinetics